CLINICAL TRIAL: NCT06662825
Title: SEG-2022-01 Patient Characteristics and Treatment Patterns From Early Crizanlizumab Use in Real-world Setting: Preliminary Analysis From Select Sickle Cell Centers
Brief Title: Real World Patient Characteristics and Treatment Patterns From Crizanlizumab Use: Preliminary Analysis From Select Sickle Cell Centers
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CSEG101AUS20
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Crizanlizumab Cohort: Patients with sickle cell disease (SCD) who had received at least one dose of crizanlizumab between 2019 and 2022.

SUMMARY:
This was a retrospective cohort study using secondary data from member sites of the National Alliance of Sickle Cell Centers (NASCC) with patients who had initiated crizanlizumab between 2019 and 2022.

ELIGIBILITY:
Inclusion criteria

* Any patient with a diagnosis of SCD based on high performance liquid chromatography (HPLC) or hemoglobin electrophoresis at treating institution.
* Treatment order for crizanlizumab; Index date was defined as the date for the first crizanlizumab treatment.
* At least 12 months of available electronic medical record (EMR) data pre-index date (baseline).
* Patients must have received at least one dose of crizanlizumab.
* For inclusion in pre/post analysis of effectiveness, patients must have received crizanlizumab for at least 12 months.

Exclusion criteria None identified.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Age at Index Date | Day 1 of Year 2
  Index date was defined as the date of the first crizanlizumab infusion
Gender at Index Date | Day 1 of Year 2
  Index date was defined as the date of the first crizanlizumab infusion
Race | Day 1 of Year 2
Ethnicity | Day 1 of Year 2
Insurance Type at Index Date | Day 1 of Year 2
  Index date was defined as the date of the first crizanlizumab infusion
Number of Patients Categorized by Comorbidity | Baseline
Number of Patients who Received Long-acting Opioid Medication Before Starting Crizanlizumab | Baseline
Number of Patients who Received Chronic Red Blood Cell Transfusion Therapy Before Starting Crizanlizumab Categorized by Duration of Therapy | Baseline
  Red blood cell transfusion therapy time intervals:
  * 0-3 months
  * 3-6 months
  * 6-12 months
  * >12 months
  * Unknown
Number of Patients who Received Chronic Red Blood Cell Transfusion Therapy After Starting Crizanlizumab Categorized by Duration of Therapy | Up to 1 year
  Red blood cell transfusion therapy time intervals:
  * 0-3 months
  * 3-6 months
  * 6-12 months
  * >12 months
  * Unknown
Number of Patients by Type of Disease Modifying Therapy (DMT) Received Pre- and Post-index Date | Up to 2 years
  Index date was defined as the date of the first crizanlizumab infusion.
  DMTs included:
  * Any SCD specific therapy
  * Hydroxyurea
  * Voxelotor
  * L-Glutamine
  * Other

SECONDARY OUTCOMES:
Number of Doses Received by Patients Who Continued and Discontinued Crizanlizumab Treatment | 1 year
Number of SCD-related Hospitalizations and Emergency Department Visits Pre- and Post-index Date | Up to 2 years
  Index date was defined as the date of the first crizanlizumab infusion.
Length of Stay of SCD-related Hospitalization Visits Pre- and Post-index Date | Up to 2 years
  Index date was defined as the date of the first crizanlizumab infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States